CLINICAL TRIAL: NCT03220906
Title: Comparison of Blood Pressure Measurements in Upper and Lower Extremities in Children Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB17-00268
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arterial line: Children undergoing surgical procedure with planned arterial cannula placement.
  Interventions: Other: Blood pressure measurement

INTERVENTIONS:
Other: Blood pressure measurement — Blood pressure will be measured in both upper and lower extremities.

SUMMARY:
There is very little information comparing non-invasive blood pressure (BP) readings obtained from upper and lower limbs, as well as comparing invasive and non-invasive blood pressures in the children under anesthesia. This study seeks to determine the correlation between the non-invasive BP measurements between upper and lower extremities and compare these measurements with the invasive BP as the standard for comparison.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1-3
* 0-10 years of age
* Undergoing surgical procedure with planned arterial cannula placement

Exclusion Criteria:

* ASA status >3
* Older than 10 years of age
* Patient unable to have BP taken on 1 upper and 1 lower extremity

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing a surgical procedure with planned arterial cannula placement at Nationwide Children's Hospital in Columbus, OH or King Fahad Medical City in Riyadh, Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Deviation >5 mmHg in MAP | 45 minutes
  Deviation >5 mmHg in MAP between one of the non-invasive measurements compared to invasive BP measurement at any point during the study.

SECONDARY OUTCOMES:
Deviation >10 mmHg | 45 minutes
  Deviation >10 mmHg between the non-invasive and invasive measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided